CLINICAL TRIAL: NCT04945694
Title: Ultrasound-Guided Bilateral Pecto-intercostal Fascial Block Versus Intravenous Fentanyl for Postoperative Pain Management After Pediatric Cardiac Surgery A Prospective, Randomized, Controlled Study
Brief Title: Pain Management of Pecto-intercostal Fascial Block Versus Intravenous Fentanyl After Pediatric Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD/ 21.04.462
Record Dates: First submitted 2021-06-13; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Pediatric Patients; Congenital Heart Surgery
MeSH Terms: interventions — Propofol; Sevoflurane; Atracurium; Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided bilateral pecto-intercostal fascial block (Experimental): Patients will receive bilateral ultrasound-guided pecto-intercostal fascial block
  Interventions: Other: Ultrasound-guided bilateral pecto-intercostal fascial block; Drug: Propofol; Drug: Sevoflurane; Drug: Atracurium; Device: ultrasound
- Intravenous fentanyl (Placebo Comparator): Patients will receive only incremental doses of intravenous fentanyl
  Interventions: Drug: Intravenous fentanyl; Drug: Propofol; Drug: Sevoflurane; Drug: Atracurium

INTERVENTIONS:
Other: Ultrasound-guided bilateral pecto-intercostal fascial block — - PATIENT IN SUPINE POSITION, SKIN WILL BE DISINFECTED, A HIGH-FREQUENCY LINEAR PROBE WILL BE PLACED PARALLEL TO LONGITUDINAL AXIS OF STERNUM ON LATERAL BORDER AND SCANNED LATERALLY TO IDENTIFY 4TH AND 5TH COSTAL CARTILAGE. THE PECTORALIS MAJOR MUSCLE (PMM), INTERNAL INTERCOSTAL MUSCLE (IIM), TRANSVERSUS THORACIS MUSCLE (TTM), RIBS, AND PLEURA WILL BE IDENTIFIED. COLOR DOPPLER ULTRASONOGRAPHY WILL BE USED TO DETERMINE PERFORATING BRANCHES OF INTERNAL THORACIC ARTERY, WHICH TRAVEL ANTERIORLY THROUGH THE ANTERIOR CHEST WALL, PIERCING THE INTERCOSTAL MUSCLE AND PMM. A 22G NEEDLE WILL BE INSERTED IN PLANE WITH PROBE, IN CAUDAL-TO-CRANIAL DIRECTION UNTIL THE TIP IS POSITIONED IN INTER- FASCIAL PLANE BETWEEN THE PMM AND IIM. NORMAL SALINE WILL BE USED TO DETERMINE CORRECT PLACEMENT OF NEEDLE TIP IN INTER-FASCIAL PLANE, AS SHOWN BY SEPARATION OF FASCIAL LAYERS THEN LOCAL ANESTHETIC WILL BE INJECTED
  Arms: Ultrasound-guided bilateral pecto-intercostal fascial block
Drug: Intravenous fentanyl — In this group, patients will receive only incremental doses of intravenous fentanyl
  Arms: Intravenous fentanyl
Drug: Propofol — Propofol anesthesia
Drug: Sevoflurane — Sevoflurane anesthesia
Drug: Atracurium — Intravenous atracurium
Device: ultrasound — ultrasound-guided block
  Arms: Ultrasound-guided bilateral pecto-intercostal fascial block

SUMMARY:
Cardiac surgical patients often experience significant postoperative pain at the median sternotomy site.

In pediatric cardiac surgery, the recommended pre bypass dose of fentanyl to blunt the hemodynamic and metabolic stress response is 25-50 µg/kg Today lower doses are often used in order to achieve early extubation at such doses there is no guarantee that the stress response is completely abolished one way to overcome this problem is the use of the local anesthetic technique Regional anesthetic techniques reduce pain for up to 24 hours after cardiac surgery in children.

Pectointercostal fascial block was first described by de la Torre in patients undergoing breast surgery. This novel technique blocks the anterior cutaneous nerve which is a branch of the intercostal nerve that gives sensory supply to the skin.

DETAILED DESCRIPTION:
The aim of the current study is to detect the effectiveness of pecto-intercostal fascial block in relieving postoperative pain in noncyanotic pediatric patients undergoing elective cardiac surgery the primary goal of this randomized study is to compare the postoperative pain score in the first postoperative 24 hours and to detect total dose of fentanyl requirements. The secondary goals are intraoperative hemodynamic stress response to surgical stimuli, analgesic consumption in the studied groups, cross-clamping and bypass time, time to extubation, intensive care length of stay, and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* On pump
* Elective repair of congenital simple left to right intracardiac shunt
* Median sternotomy

Exclusion Criteria:

* Refusal of their guardians
* Redo cardiac surgery
* Previous back injury
* Previous back surgery
* Kyphoscoliosis
* Local infection of the skin and subcutaneous tissue at the site of needle puncture
* Hypersensitivity to local anesthetics
* Coagulation disorders
* Renal disease
* Hepatic disease
* Pulmonary disease
* Heart failure
* Moderate to severe pulmonary hypertension.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain assessment | Postoperative day 1
  Postoperative pain will be assessed using the modified objective pain score (OPDS) in children.
Total dose of fentanyl requirements | intraoperative and 24 hrs postoperatively
  Total dose of fentanyl requirements

SECONDARY OUTCOMES:
Serum cortisol levels | Basal and one-hour postoperatively
Heart rate [HR] | before induction of anesthesia (basal value), after induction of anesthesia, after skin incision, after sternotomy, 15 min after CPB and after the closure of sternum
Invasive mean arterial blood pressure [MAP] | before induction of anesthesia (basal value), after induction of anesthesia, after skin incision, after sternotomy, 15 min after CPB and after the closure of sternum

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Ghanem, MD, Study Director — Assistant professor, MD anesthesia Department, Faculty of Medicine, Mansoura University, Egypt; Enas Abd Elmotlb, MD, Study Chair — professor, MD anesthesia Department, Faculty of Medicine, Mansoura University, Egypt
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De -identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: will be available within 6 months of study completion
Access Criteria: data access requests will be reviewed by an external independent review panel .requestors will be required to sign a data access agreement